CLINICAL TRIAL: NCT04463550
Title: GFAP Auto-immunity : a French Cohort Study
Acronym: GFAP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: GFAP
Record Dates: First submitted 2020-04-17; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-06

CONDITIONS: Autoimmune GFAP Astrocytopathy
Keywords: Acidic Protein IgG; astrocytopathy; meningoencephalomyelitis; perivascular-radial parenchymal enhancement; autoimmune; paraneoplasic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients GFAP-IgG positive in serum and/or CSF: Patients developing clinical autoimmune encephalitis or meningoencephalomyelitis with anti-GFAP antibodies, managed by the National Reference Center for Paraneoplastic Syndromes and Autoimmune Encephalitis or the National Reference Center for Centre de référence for Neuro-inflammatory diseases of the brain and the spinal cord at the Neurological Hospital of Bron.
  Interventions: Other: Description and analysis

INTERVENTIONS:
Other: Description and analysis — Retrospective, non-interventional study, using clinical, biological, radiological and therapeutic data collected during the initial diagnosis and follow-up.

SUMMARY:
Glial fibrillary acidic protein (GFAP)-Immunoglobulin G (IgG) have recently been described as a biomarker of a novel inflammatory central nervous system (CNS) disorder, termed autoimmune GFAP astrocytopathy. Thus far, four major clinical series have been published (two from Mayo Clinic USA, one from Italy and one from China). GFAP-IgG detected in serum or in cerebrospinal fluid, by tissue-based assay and confirmed by cell-based assay, are associated with encephalitis or meningoencephalitis of acute or subacute onset, less frequently with myelitis or optic disk edema. The characteristic MRI feature is brain linear perivascular radial gadolinium enhancement in the white matter perpendicular to the ventricle, consistent with the immunohistochemical staining pattern of GFAP in rodent brain sections. Approximately 20% of reported cases are associated with a neoplasm (ovarian teratoma mostly). Coexisting neural autoantibodies are described in some patients, N-methyl-D-aspartate (NMDA)-receptor (R)-IgG mostly, followed by aquaporin 4 (AQP4)-IgG. The disease is usually corticosteroid responsive although relapse can occur. In contrast, Chinese patients display poorer outcomes. Pathophysiology is not well understood but the intracellular antigen location makes GFAP-IgG unlikely pathogenic whereas animal models and neuropathologic data suggest a T-cell immune-mediated disorder.

The aim of the investigators is to report the first French cohort of patients GFAP-IgG positive. Investigators retrospectively assessed clinical, immunological and radiological features, treatment response and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Positive GFAP-Ab in serum and/or CSF tested by immunohistochemistry on mouse brain slices and confirmed by cell-based assay (CBA) of HEK293 cells expressing GFAP.
* Diagnosis and follow-up in France
* No age limit : from 0 to unlimited age

Exclusion Criteria:

* Patients GFAP-IgG negative in serum and CSF
* Absence of complete clinicopathological data
* Foreign follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients GFAP-IgG positive in serum and/or CSF
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Report retrospectively clinical data of patients GFAP-IgG positive. | 13 months
  Describe prodromes (yes or no), neurologic signs and clinical course (acute/subacute - yes or
  no - or progressive onset - yes or no), if admitted in intensive care units (yes or no), retrospectively provided by
  the treating physicians using a structured questionnaire.or progressive onset), if admitted in intensive care units, neoplastic and dysimmune associated diseases and T cell dysregulation condition .

SECONDARY OUTCOMES:
Describe GFAP-antibody test results. | 13 months
  positivity of GFAP α -IgG in cerebrospinal fluid, in serum and isoform type at diagnostic and follow up.
  positivity of GFAP α -IgG in cerebrospinal fluid, in serum and isoform type at diagnostic and follow up.
demographic data of patients GFAP-IgG positive : age at onset | 13 months
  age at onset (years) retrospectively provided by the treating
  physicians using a structured questionnaire

OTHER OUTCOMES:
demographic data of patients GFAP-IgG positive : phenotype | 13 months
  Report if caucasian (yes or no) retrospectively provided by the treating
  physicians using a structured questionnaire
demographic data of patients GFAP-IgG positive : sex | 13 months
  Report if female sex (yes or no) retrospectively provided by the treating
  physicians using a structured questionnaire
  physicians using a structured questionnaire
associated conditions of patients GFAP-IgG positive | 13 months
  Report if neoplastic and dysimmune associated diseases and T cell dysregulation condition (yes or no)
  physicians using a structured questionnaire
  physicians using a structured questionnaire
Report cerebrospinal fluid white cell count | 13 months
  white cell count (/mm3)
Report cerebrospinal fluid protein level | 13 months
  protein level (g/L)
Report cerebrospinal fluid glucose level | 13 months
  glucose level (mmol/L)
Report number of oligoclonal bands in cerebrospinal fluid | 13 months
  number of oligoclonal bands
Describe MRI features. | 13 months
  Head and medullar MRI at diagnostic and follow up were reviewed by a neuroradiologist. scale) at each relapse and last follow up.
Report other paraclinic findings : electroencephalographic results. | 13 months
  Describe electroencephalographic results at diagnostic and follow up when done .
Report other paraclinic findings : electromyographic results. | 13 months
  Describe electromyographic results at diagnostic and follow up when done .
Report ophthalmic exam : visual acuity | 13 months
  Describe visual acuity (/10) at diagnostic and follow up when done .
Report ophthalmic exam : ocular fundus. | 13 months
  Describe ocular fundus at diagnostic and follow up results when done .
Report ophthalmic exam : visual field. | 13 months
  Describe visual field at diagnostic and follow up when done .
Report ophthalmic exam : optical coherence tomography. | 13 months
  Describe optical coherence tomography (RNFL thickness) at diagnostic and follow up when done .
Report histologic findings. | 13 months
  Describe histologic results at diagnostic and follow up when done .
Report treatments and response. | 13 months
  Describe acute and long-term treatments administered and response.
Report outcome. | 13 months
  Describe outcome (modified Rankin scale) at each relapse and last follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Romain MARIGNIER, Study Director — Centre de référence des maladies inflammatoires rares du cerveau et de la moelle, Lyon, France
Locations (1):
- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No